CLINICAL TRIAL: NCT02950519
Title: Assessing Endotracheal Tube Cuff Pressures in Mechanically Ventilated Patients
Brief Title: Endotracheal Tube Cuff Pressures in Ventilated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barnes-Jewish Hospital (Other)
Responsible Party: Principal Investigator, Peggy Watts, MS, Barnes-Jewish Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201605155
Record Dates: First submitted 2016-10-06; First posted 2016-11-01 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Pneumonia, Ventilator-Associated
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- As needed Cuff Pressure Checks (Active Comparator): Cuff pressure checks upon intubation and after any manipulation of ET tube
  Interventions: Other: monitoring of cuff pressures
- Cuff Pressure checks every 8 hrs (Experimental): Cuff pressure checks upon intubation, after manipulation of ET tube, and minimum of 8 hr interval
  Interventions: Other: monitoring of cuff pressures

INTERVENTIONS:
Other: monitoring of cuff pressures — Cuff pressure will be checked per standard and additionally a minimum of every 8 hours.

SUMMARY:
There is no accepted standard for the frequency of monitoring endotracheal tube cuff pressures (ETCP). Investigators plan on comparing two strategies for monitoring ETCP in mechanically ventilated patients. The two strategies will be the currently employed practice at Barnes-Jewish Hospital (BJH) which requires ETCP to be assessed immediately after the endotracheal tube is placed and after any manipulation of the endotracheal tube to include repositioning, manipulation of the cuff volume, or presence of an audible leak. Investigator will compare this current practice to a more intensive monitoring of ETCP which is employed at some hospitals and includes the same elements as noted in the current practice plus monitoring ETCP every work shift (every 8 hours or three times per day).

DETAILED DESCRIPTION:
There is no accepted standard for the frequency of monitoring endotracheal tube cuff pressures (ETCP). Investigator plans on comparing two strategies for monitoring ETCP in mechanically ventilated patients. The two strategies will be the currently employed practice at Barnes-Jewish Hospital (BJH) which requires ETCP to be assessed immediately after the endotracheal tube is placed and after any manipulation of the endotracheal tube to include repositioning, manipulation of the cuff volume, or presence of an audible leak. The alternate practice will be pre-scheduled as is performed at other hospitals and includes the same elements as noted in the current practice but also require monitoring ETCP a minimum of every work shift (every 8 hours or three times per day). The ETCP will be assessed using a standard manometer. The two practices will be compared by assessing patients assigned to odd and even beds in the medical ICU (8400 ICU) with alternate methods. Specifically, patients in odd numbered rooms will have ETCP checked per the current Barnes-Jewish practice and those in even rooms having the additional checks of ETCP performed immediately following intubation as well as every shift and when when assessed required by respiratory therapist. It is important to note that the respiratory therapists performing ETCP assessments are simply performing a routine 2- 3 minute task (per cuff pressure measurement) while taking care of patients on mechanical ventilation.

Our hypothesis is that increased monitoring frequency of ETCP will not result in a decrease in the duration of mechanical ventilation for patients admitted to the medical intensive care unit (ICU) of BJH or a reduction in ventilator-associated events.

Currently there is no accepted gold standard for the frequency of monitoring ETCP. There are widely different strategies reported for monitoring ETCP to include continuous monitoring. The goal of ETCP monitoring is to maintain the ETCP between 20-30 cmH2O in order to minimize cuff leaks and pressure injury to the tracheal mucosa. It is known that 20 to 30% of the time the ETCP may deviate above or below this threshold. However, the impact of such deviation on clinical outcomes is not well described in the medical literature. The two most common methods for assessing ETCP is the use of a manometer and/or setting a minimal leak, with the former being the most accepted method. However, the optimal frequency for conducting manometric monitoring of ETCP is unknown. One recent study suggests that the act of measuring ETCP frequently in order to achieve a desired pressure level results in the removal of air from the cuff and can result in under inflation of the cuff. However, a recent animal study suggests that the material used to manufacture the endotracheal tube cuff may play a more important role in determining the presence or absence of mucosal injury, with polyurethane being better than polyvinylchloride. The main problem with these studies is the failure to assess clinical outcomes at the bedside with the use of various strategies to maintain an appropriate endotracheal tube cuff seal. A recent survey of intensivists in Queensland Australia and accompanying systematic literature review made the following conclusions regarding ETCP monitoring: "Twenty-eight out of twenty-nine respondents reported routinely monitoring tracheal cuff function, primarily employing cuff pressure measurement (26/28). Target cuff pressures varied, with 3/26 respondents aiming for 10 to 20 cmH2O, 10/26 for 21 to 25 cmH2O, and 13/26 for 26 to 30 cmH2O. Fifteen out of twenty-nine reported they had no current guideline or protocol for tracheal cuff management and only 16/29 indicated there was a dedicated area in the clinical record for reporting cuff intervention. The results indicated that many ICUs across Queensland routinely measure tracheal cuff function, with most utilising pressure monitoring devices. Consistent with existing literature, the optimum cuff pressure remains uncertain. Most, however, considered that this should be a routine part of ICU care". Thus, the available literature on ETCP and their relationship to clinical outcomes is lacking.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated patients intubated in a medical intensive care unit

Exclusion Criteria:

* Patient requiring prone positioning, lung transplant and neutropenic patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2016-10; Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Ventilator Associated Condition (VAC) as defined by CDC | 48 hours after intubation
  Lung Condition that developed in association with mechanical ventilation

SECONDARY OUTCOMES:
Length of stay (hospital) | Time in days of hospital stay for patients admitted and discharged for a period up to 6 months
  Through hospital admission until hospital discharge for patients admitted and discharged for a period up to 6 months
Hospital mortality | Any time during hospitalization up to a period of 6 months
  Through hospital admission until hospital discharge up to a period of 6 months
Ventilator Associated Pneumonia (VAP) | 48 hrs after intubation
  Pneumonia that developed in association with mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Marin Kollef, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes-Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided
We are undecided on this point.